CLINICAL TRIAL: NCT06637579
Title: Effects of Universal Exercise Unit Therapy With Task-oriented Training on Lower Extremity Gross Motor Function and Balance in Cerebral Palsy Children
Brief Title: Effects of Universal Exercise Unit Therapy With Task-oriented Training in CP Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/24/0210
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Cerebral Palsy Children

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Group A received universal exercise unit therapy with task-oriented strength training.
  Interventions: Other: universal exercise unit therapy with task oriented strength training
- Group B (Experimental): Group B received task-oriented training for gross motor functioning.
  Interventions: Other: Task-oriented training for gross motor functioning

INTERVENTIONS:
Other: universal exercise unit therapy with task oriented strength training — Leg press, Sit to stand, Half knee rise, Lateral step up, Forward step up.
  Arms: Group A
Other: Task-oriented training for gross motor functioning — Standing transfer (hip abduction/adduction), Stair climbing (hip extension, calf raise), Walking and gait training, Reaching and grasping activities.
  Arms: Group B

SUMMARY:
Cerebral palsy is a problem that affects the development and motor skills caused by early non-progressive central nervous system damage. Muscle rigidity, spasticity, fragility, uncontrolled movement, or a combination of these abnormalities characterized it. Therapeutic usage of the universal exercise unit is common. Also called a spider cage or monkey cage. This device helps people with motor problems, especially cerebral palsy. This metal 3-dimensional contraption uses wires, rubber bands, pulleys, weights, and belts. The goal is to engage the vestibular and proprioceptive systems, which are necessary for balance, coordination, and awareness.

DETAILED DESCRIPTION:
A Randomized Clinical Trial (RCT) design will be employed, conducted at the Sialkot Medical and Physiotherapy Center over 10 months following synopsis approval. The anticipated sample size, accounting for a 20% attrition rate, will be 34 participants in each of the two study groups. Group A will undergo Universal Exercise Unit (UEU) therapy along with task oriented training, while Group B will receive task-oriented training for gross motor functioning. The sampling technique will be Non-probability convenience sampling, with inclusion criteria comprising children aged 5-15 diagnosed with spastic cerebral palsy, of both genders and in stable health condition. The data collection tools include the Gross Motor Function Measure 88 (GMFM 88), Trunk Impairment Scale (TIS) and pediatric balance scale. The analysis will be conducted using SPSS for Windows software version 25. Training sessions, lasting 6 weeks, will be conducted twice a week, and data will be collected before and after each session. The UEU therapy will focus on various movements facilitated by the equipment, while the task-oriented training will be personalized, targeting specific functional limitations through activities simulating daily tasks.

ELIGIBILITY:
Inclusion Criteria:

* Children who were spastic and able to understand and follow commands. Children aged 5-15 years old. Gross Motor Function Classification System (GMFCS) level I-III. Youngsters are capable of walking and standing on their own.

Exclusion Criteria:

* Children with severe physical limitations and disabilities. Children with planned surgeries in the next 6 months. Any musculoskeletal or orthopedic conditions limiting participation in exercise programs.

Kids with planned surgical or medical surgeries during the study period. Children with impaired cognition. Children with hearing impairment and visual impairment.

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
GMFM 88 (gross motor function measure) | 6 weeks
  GMFM is an assessment tool used to evaluate and measure gross motor function in CP
TIS (trunk impairment scale) | 6 weeks
  TIS is a clinical assessment tool designed to evaluate trunk control
Pediatric Berg Balance Scale | 6 weeks
  The Pediatric Balance Scale is used to assess functional balance skills in school-aged children

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Asrar Yousaf, M.phil, Principal Investigator — Riphah International University
Locations (1):
- Sialkot Medical and Physiotherapy Center, Sialkot, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No